CLINICAL TRIAL: NCT01474278
Title: A Multi-centre, Randomized, Double-blind, Placebo-controlled, Two-period Cross-over, Exploratory Biomarker and Safety and Tolerability Study of a Single Dose of RO5028442 in Adult Male High-functioning Autistic Patients
Brief Title: A Study of RO5028442 in Adult Male High-Functioning Autistic Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: BP27801
Record Dates: First submitted 2011-11-15; First posted 2011-11-18 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Autistic Disorder
MeSH Terms: conditions — Autistic Disorder | interventions — (6-chloro-1-(2-(dimethylamino)ethyl)indol-3-yl)-spiro(1H-isobenzofuran-3,4'-piperidine)-1'-yl-methanone

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: RO5028442
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Single dose
  Arms: 2
Drug: RO5028442 — Single dose
  Arms: 1

SUMMARY:
This multi-center, randomized, double-blind study will evaluate exploratory biomarkers and the safety and tolerability of a single dose of RO5028442 in adult male high-functioning autistic patients. In a cross-over design, patients will be randomized to receive either a single dose of RO5028442 or matching placebo with a washout period of 7-14 days. Anticipated time on study is up to approximately 9 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of Autistic Disorder as defined by DSM-IV, confirmed by the team and supported with the Autistic Diagnostic Observation Schedule (ADOS)
* Male adults, 18 to 45 years of age
* IQ > 70 (Wechsler Adult Intelligence Scale-Full scale)
* Body mass index (BMI) 18 to 35 kg/m2 inclusive
* Aberrant Behavior Checklist (ABC) - Irritability subscale score </= 13

Exclusion Criteria:

* Positive urine test for drugs of abuse
* Alcohol and/or substance abuse/dependence during the last 12 months
* Positive for hepatitis B, hepatitis C or HIV infection
* Clinically relevant cardiovascular, renal, hepatic or hematologic disease or disorder
* Active inflammatory pulmonary disease
* History of epilepsy/seizure disorder (except for simple febrile seizures)
* Initiation of new or major change in psychosocial intervention within 4 weeks prior to randomization
* Treatment with any investigational agent within 90 days prior to screening
* History of hypersensitivity or allergic reactions

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2011-12; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Efficacy: Behavior assessments | up to 24 hours post-dose
Safety: Incidence of adverse events | up to 24 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (3):
- United States (3):
  - Los Ageles, California
  - New Haven, Connecticut
  - The Bronx, New York

REFERENCES:
- [Derived] Umbricht D, Del Valle Rubido M, Hollander E, McCracken JT, Shic F, Scahill L, Noeldeke J, Boak L, Khwaja O, Squassante L, Grundschober C, Kletzl H, Fontoura P. A Single Dose, Randomized, Controlled Proof-Of-Mechanism Study of a Novel Vasopressin 1a Receptor Antagonist (RG7713) in High-Functioning Adults with Autism Spectrum Disorder. Neuropsychopharmacology. 2017 Aug;42(9):1914-1923. doi: 10.1038/npp.2016.232. Epub 2016 Oct 6. PMID 27711048